CLINICAL TRIAL: NCT02064257
Title: The Listening Project: Tuning Into Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Australian Childhood Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-2304
Record Dates: First submitted 2014-02-10; First posted 2014-02-17 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Auditory Perceptual Disorders; Stress Disorder
Keywords: autonomic nervous system; auditory processing disorder; social behavior
MeSH Terms: conditions — Auditory Perceptual Disorders; Stress Disorders, Traumatic; Social Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Participants will be included in all pre-intervention and post-assessment measures. Participants will receive the Listening Project Protocol intervention. The duration of the intervention is approximately 45 minutes per day, for 5 consecutive days.
  Interventions: Behavioral: Listening Project Protocol
- Assessment-only group (No Intervention): The assessment-only group will participate in all pre- and post-intervention assessments, but will not receive the Listening Project Protocol.

INTERVENTIONS:
Behavioral: Listening Project Protocol — The intervention will consist of listening to computer-altered acoustic stimulation, designed to modulate the frequency band of vocal music passed to the participant. The frequency characteristics of the acoustic stimulation are selected to emphasize the relative importance of specific frequencies in conveying the information embedded in human speech. Modulation of the acoustic energy within the frequencies of human voice, similar to an exaggerated vocal prosody, are hypothesized to recruit and modulate the neural regulation of the middle ear muscles and to functionally reduce sound hypersensitivities and improve auditory processing.
  Arms: Intervention group

SUMMARY:
A research project funded by the Australian Childhood Foundation (ACF) will be conducted in Australian facilities of the ACF to evaluate the effectiveness of the Listening Project Protocol (LPP) in children with a trauma history. The LPP is designed as a "neural exercise" to reduce auditory hypersensitivities, to improve auditory processing of speech, and to improve behavioral state regulation. The LPP uses acoustic stimulation to exercise the neural regulation of the middle ear structures to rehabilitate and to normalize the acoustic transfer function of the middle ear structures. The current study is being conducted to evaluate efficacy and feasibility of the LPP and will use objective measures to evaluate changes in acoustic transfer function of the middle ears structures, auditory processing skills, physiological state regulation, and sensory symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Children must be between ages 7-14 years
* Children and parent providing permission must be able to read/speak in English
* Children must be receiving services from the Child Trauma Service unit of the Australian Childhood Foundation

Exclusion Criteria:

* Children who wear a hearing-device
* Children with a history of heart disease
* Children who are currently being treated for seizure disorder

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Auditory hypersensitivity | pre-intervention (within 1 week before intervention), post-intervention (within 1 week after intervention), 1 month post-intervention
  Brain-Body Center Sensory Scales (BBC Sensory Scales) (parental questionnaire)

SECONDARY OUTCOMES:
Autonomic state regulation | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 1 month post-intervention
  heart rate, heart period, high-frequency heart rate variability/respiratory sinus arrhythmia
Auditory processing | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 1 month post-intervention
  filtered words, competing words subscales of SCAN
social behavior | post-intervention (within 1 week after the intervention), 1 month post-intervention
  Listening Project Parent Questionnaire
Middle ear muscle transfer function | pre-intervention (within 1 week before intervention), immediate post-intervention (within 1 week after intervention), 1 month post-intervention
  MESAS (Middle Ear Sound Absorption System)

CONTACTS AND LOCATIONS:
Overall Officials: Keri J Heilman, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Child Trauma Service Unit, Australian Childhood Foundation, Ringwood, Victoria, Australia